CLINICAL TRIAL: NCT01109810
Title: Immunoglobulin, Diagnosis, Evaluation, and Key Learnings Patient Registry (IDEaL™)
Acronym: IDEaL
Status: Completed | Type: Observational
Sponsor: Coram Clinical Trials (Other)
Responsible Party: Sponsor
Other Study IDs: CT-10-02
Record Dates: First submitted 2010-04-21; First posted 2010-04-23 (Estimated); Last update posted 2022-06-22 (Actual); Status verified 2022-06

CONDITIONS: IVIg or SCIg Therapy in the Home or at Alternate Site

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- IVIg and SCIg therapy: Patients receiving Ig therapy by IV or SC route in the home or alternate site setting

SUMMARY:
The IDEaL registry is a cooperative, observational registry focused on immunoglobulin use in the U.S. The registry is a deliberate and purposeful assembly of clinical and humanistic knowledge that is intended to act as a longitudinal database, tracking outcomes of routine clinical practice.

The central goal of the registry is to provide a mechanism that allows for a better understanding of how immunoglobulin therapy is being used in a real-world clinical setting. The data gathered will help the industry gain a better understanding surrounding the therapeutic value of immunoglobulin therapy and subsequently improve practices, reduce medical costs, and ultimately improve the clinical outcomes for the patients receiving immunoglobulin therapy

DETAILED DESCRIPTION:
The registry's goal is to significantly contribute to the medical understanding of Ig therapy and to improve the quality of care for patients receiving Ig therapy in the United States through active publication of registry findings and disease management approaches.

The IDEaL program represents a unique and powerful method for the collection of:

Patient Level / Humanistic Data / Quality of Life Physician Level / Practice Patterns Clinical Data / Therapeutic Outcomes Reimbursement / Impact on Treatment / Policy Decisions

Whereby:

Accelerating innovation Producing faster knowledge gains Improving awareness of patient outcomes and disease burden Providing a clearer understanding of therapy impact on patients' quality of life.

The objectives of the Registry are:

to enhance the understanding of the variability, progression, and natural history of disease requiring Ig therapy with the ultimate goal of better guiding and assessing therapeutic intervention; to provide the Ig medical community with recommendations for monitoring patients and to provide reports on patient outcomes to help optimize patient care; and to serve as an active knowledge base that can provide population-management information, which can be used to generate patient-management and practice-management tools; and

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Any age, disease, or gender requiring Ig therapy
* Agree to the use of Coram's infusion services after entry into IDEaL Registry

Exclusion Criteria:

* Unable to start, or stops taking Ig therapy
* Use of an insurance provider for which Coram's services are not covered/authorized.
* Have previously participated in the IDEaL Registry and revoked consent to use their PHI

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The IDEaL Registry program will collect data representative of patients receiving Ig therapy (IVIg and SCIg) in a homecare setting and/or through Coram's ambulatory infusion suites.
Sampling Method: Non-Probability Sample
Enrollment: 496 (Actual)
Dates: Start 2010-09-08 (Actual); Primary Completion 2022-06-10 (Actual); Study Completion 2022-06-10 (Actual)

PRIMARY OUTCOMES:
Disease by geographic region (and/or Investigative Site), age, therapeutic indication (immunologic/neurologic) | Baseline
  Recorded from referral form
Infection incidence by route, dose, and age | every 6 months
  Infection incidence, route, dose recorded from Clinical Progress reports Immune Replacement Efficacy section

SECONDARY OUTCOMES:
Dosing information by disease type, Investigative Site, and therapeutic indication | Estimated for baseline and 1 year
  Dosing collected from Clinical Progress Reports and/or Medication Record
Adverse events and serious adverse events by disease type and relation to Ig therapy | Estimated for baseline and 1 year
  Collected from Clinical Progress Reports Therapy Tolerance section
IVIg vs SCIg by disease type and geographic region (and/or investigative site) | Baseline
  Route collected from Clinical Progress Reports and/or Medication Record
Current state of disease by number of Ig doses received and overall | Estimated for 1 year
  Ig doses monitored by missed dose section of Clinical Progress Report and Shipping Records
Payor type by investigator site | Estimated for baseline and 1 year
  Recorded from referral information
Insurance reimbursement issues | Estimated for baseline and 1 year
  Obtained when patient has to discharge from study due to insurance change and Coram not a provider
Concomitant medication use by disease type and therapeutic indication | Estimated for baseline and 1 year
  Collected from Medication Record

CONTACTS AND LOCATIONS:
Overall Officials: Luqman Seidu, MD, Principal Investigator — Omni Allergy, Immunology, and Asthma
Locations (1):
- Coram Clinical Trials, Centennial, Colorado, United States

REFERENCES:
- [Background] IMMUNOGLOBULIN THERAPY AND QUALITY OF LIFE IN PRIMARY IMMUNODEFICIENCY PATIENTS WITH NON-INFECTIOUS PULMONARY COMPLICATIONS Checkley, A. et al. Annals of Allergy, Asthma & Immunology , Volume 121 , Issue 5 , S9 - S10
- [Result] Kearns S, Kristofek L, Bolgar W, Seidu L, Kile S. Clinical Profile, Dosing, and Quality-of-Life Outcomes in Primary Immune Deficiency Patients Treated at Home with Immunoglobulin G: Data from the IDEaL Patient Registry. J Manag Care Spec Pharm. 2017 Apr;23(4):400-406. doi: 10.18553/jmcp.2017.23.4.400. PMID 28345437
- [Result] P259 Optimizing subcutaneous dosing of immunoglobulin in obese primary immune deficiency patients treated in the home Checkley, A. et al. Annals of Allergy, Asthma & Immunology , Volume 119 , Issue 5 , S65